CLINICAL TRIAL: NCT04609449
Title: A Comparison Between Short vs. Long Biliopancreatic Limb Gastric Bypass: Early Outcomes of a Prospective Study
Brief Title: A Comparison Between Short vs. Long Biliopancreatic Limb Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CARLOS ZERRWECK LOPEZ (Other Government)
Responsible Party: Sponsor-Investigator, CARLOS ZERRWECK LOPEZ, Professor and Head of Department., Hospital General Tlahuac
Organization: Hospital General Tlahuac (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZL-030619
Record Dates: First submitted 2020-06-15; First posted 2020-10-30 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Bariatric Surgery; Metabolic Surgery; Roux-en-Y Gastric Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long biliopancreatic limb (Experimental): Patients submitted to long biliopancreatic limb Roux-en-Y gastric bypass.
  Interventions: Procedure: Long biliopancreatic limb Roux-en-Y gastric bypass.
- Standard biliopancreatic limb (Active Comparator): Patients submitted to standard Roux-en-Y gastric bypass.
  Interventions: Procedure: Standard Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Long biliopancreatic limb Roux-en-Y gastric bypass. — Long biliopancreatic limb Roux-en-Y gastric bypass.
  Arms: Long biliopancreatic limb
Procedure: Standard Roux-en-Y gastric bypass — Standard Roux-en-Y gastric bypass
  Arms: Standard biliopancreatic limb

SUMMARY:
Prospective study including patients submitted to RYGB (n=94) and L-RYGB (n=94) at a single institution. The aim was to compare the effect on comorbidities and weight loss of a long biliopancreatic limb Roux-en-Y gastric bypass (L-RYGB), compared with a standard RYGB. Procedure selection was randomly assigned (1:1), and surgeries were performed, during 24 months (2016-2017). Weight loss, comorbidities control and nutritional status were assessed at baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient submitted to bariatric surgery
* All patients met the guidelines defined by the National Institutes of Health (NIH) consensus: BMI equal or greater to 40kg/m2 or BMI 35 - 40 kg/m2 with some comorbidity

Exclusion Criteria:

•Patients with incomplete surgery data sheet and those submitted to other type of bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months
  Measures: Weight in kilograms
Weight loss | 12 months
  Measures: Body Mass Index
Weight loss | 12 months
  Measures: Percent of excess weight loss
Weight loss | 12 months
  Measures: Percent of total weight loss

SECONDARY OUTCOMES:
Complete Diabetes Remission Rate | 12 months
  Measures: No need for anti-diabetics while on glucose <100 mg/dl and HbA1c% <6
Major early complications | First 30 days
  Measure: Rate of re-operations and re-admissions
Major late complications | 2-12 months
  Measure: Rate of re-operations and re-admisions
Nutritional status | 12 months
  Measure: serum albumin (gr/dL)
Nutritional status | 12 months
  Measure: serum total proteins (gr/dL)
Nutritional status | 12 months
  Measure: hemoglobin (g/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Zerrweck, MD, Study Director — Head of Department. The Obesity Clinic at Hospital General Tlahuac; Antonio Herrera, MD, Principal Investigator — The Obesity Clinic at Hospital General Tlahuac
Locations (1):
- Hospital General Tlahuac, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No